CLINICAL TRIAL: NCT06911775
Title: Exploring Inflammatory and Regulatory Eosinophil Subpopulations: the Path to Precision Medicine for the Treatment of Eosinophilic-associated Diseases
Brief Title: Eosinophil Subpopulations in Eosinophilic-associated Diseases
Acronym: IREOS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Alessandra Vultaggio, Principal investigator, researcher, University of Florence
Other Study IDs: 26188-OSS
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Eosinophilic Asthma; Eosinophilic Granulomatosis With Polyangiitis (EGPA); Hypereosinophilic Syndrome (HES)
Keywords: Eosinophils; EGPA; HES; EA; Eosinophilic asthma; Eosinophil subpopulations; Flowcytometry; Biomarker; Asthma severity; EGPA severity
MeSH Terms: conditions — Pulmonary Eosinophilia; Churg-Strauss Syndrome; Hypereosinophilic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy donors: 25 healthy subject
- EA: 80 eosinophilic asthma patients
- EGPA: 30 EGPA patients
- HES: 25 HES patients

SUMMARY:
This single-center, non-commercial study will involve 160 participants (80 with eosinophilic asthma (EA), 30 with eosinophilic granulomatosis with polyangiitis (EGPA), 25 with hypereosinophilic syndrome (HES), and 25 healthy donors) to investigate eosinophil subpopulations in these diseases. The study will run from Q4 2024 to Q4 2026.

Objectives:

Primary: To verify two eosinophil subpopulations (iEos and rEos) in EGPA and HES and analyze the role of type 2 cytokines on their plasticity.

Secondary: Compare iEos proportion between different eosinophilic diseases and correlate with disease severity.

Exploratory: Assess the effect of mepolizumab on eosinophil subpopulations in vitro.

Population: Adults aged 18-75 with EA, EGPA, or HES, and healthy controls. EA patients must have >300 eosinophils/mcL, EGPA requires asthma + eosinophilia + other specific features, and HES requires high eosinophil counts (>1500 cells/mL).

Methods: Data will be analyzed using Mann-Whitney U, ANOVA, and Spearman correlation tests, with results presented as mean ± SEM.

This study will help explore eosinophil behavior in eosinophilic diseases and evaluate mepolizumab's effects on these cells.

DETAILED DESCRIPTION:
Introduction Eosinophils (Eos) play a crucial role in both normal physiological functions and various pathological conditions. They are primarily recognized for their involvement in immune defense against infections, including parasitic, bacterial, and viral infections, as well as in cancer surveillance. However, they are also key contributors to eosinophil-associated diseases (EADs) such as bronchial asthma, chronic rhinosinusitis with nasal polyps (CRSwNP), eosinophilic granulomatosis with polyangiitis (EGPA), and hypereosinophilic syndrome (HES).

Recent research has revealed that eosinophils exist in distinct subpopulations with unique phenotypic characteristics and functions. These subpopulations, referred to as resident eosinophils (rEos) and inflammatory eosinophils (iEos), have been primarily studied in healthy tissues and in conditions like severe eosinophilic asthma (SEA) and CRSwNP. While rEos are believed to contribute to tissue homeostasis and immune regulation, iEos are associated with inflammatory responses. Studies in mouse models have demonstrated the presence of these subpopulations in lung tissue, but their role in human disease remains less understood.

Although there is emerging evidence suggesting the presence of these eosinophil subsets in human peripheral blood and nasal polyp tissue, they have not been fully characterized in other EADs such as EGPA and HES. Understanding whether these subpopulations exist in these diseases and how they are influenced by type 2 cytokines could provide valuable insights into disease mechanisms. Furthermore, as eosinophil-targeted therapies such as Mepolizumab (an anti-IL-5 monoclonal antibody) are already in clinical use, clarifying their specific effects on these eosinophil subsets could help optimize treatment strategies.

Study Rationale and Objectives This study aims to expand on previous findings by investigating whether distinct eosinophil subpopulations exist in EGPA and HES patients. Additionally, the study seeks to analyze how type 2 cytokines influence the differentiation and function of these eosinophil subsets. A key aspect of this research is assessing the effect of Mepolizumab on rEos and iEos, particularly whether it selectively targets inflammatory eosinophils without affecting homeostatic eosinophils.

The primary objectives of this study include:

Confirming the presence of two distinct eosinophil subpopulations in EGPA and HES.

Investigating the impact of type 2 cytokines on eosinophil plasticity and function.

Secondary objectives involve comparing iEos proportions across different eosinophilic diseases and analyzing their correlation with disease severity. Additionally, the study will explore how in vitro exposure to Mepolizumab affects the balance between rEos and iEos in EGPA and HES patients.

Study Design The study will involve patients diagnosed with severe eosinophilic asthma (SEA), EGPA, and HES, along with a control group of healthy donors. Blood samples will be collected and analyzed using flow cytometry to characterize eosinophil subpopulations. In vitro experiments will assess the effects of type 2 cytokines (such as IL-5, IL-3, GM-CSF, IL-4, and IL-13) on these eosinophil subsets, as well as the impact of Mepolizumab.

Subject Selection and Eligibility Criteria Participants must be between 18 and 75 years old and diagnosed with SEA, EGPA, or HES. Healthy donors within the same age range will be included as controls. Individuals with chronic lung diseases (such as COPD), other immune-mediated inflammatory conditions, recent infections, parasitic infestations, or immunosuppressive treatments will be excluded to ensure a clear focus on eosinophilic-driven inflammation.

Ethical Considerations and Study Management This study will adhere to ethical guidelines outlined in the Declaration of Helsinki and Good Clinical Practice (GCP) regulations. Informed consent will be obtained from all participants, ensuring they fully understand the study's purpose and procedures. Ethical approval will be secured from the relevant institutional review boards before the study commences.

Biological samples will not be stored beyond their immediate use, and strict chain-of-custody procedures will be followed. If a participant withdraws consent, their samples will be immediately destroyed unless they have already been analyzed.

Statistical Analysis and Expected Outcomes This is an exploratory pilot study, and an estimated 135 patients (80 SEA, 30 EGPA, 25 HES) and 25 healthy donors will be recruited. Statistical methods, including Mann-Whitney U tests, ANOVA, and Spearman correlation tests, will be used to analyze the data. The primary focus will be to determine the proportion of iEos and rEos in different disease states and evaluate their response to cytokine stimulation and Mepolizumab treatment.

If successful, this study could lead to a deeper understanding of eosinophil biology and its implications in eosinophilic disorders. More importantly, it could refine therapeutic strategies by identifying whether Mepolizumab specifically targets inflammatory eosinophils while preserving homeostatic ones, ultimately leading to more personalized treatment approaches for patients with EADs.

ELIGIBILITY:
Inclusion Criteria:

- For inclusion in the study subjects should fulfill the following criteria based on local regulations:

Patients with Asthma, or EGPA or HES:

1. Age between 18 and 75 years at the time of signing the informed consent
2. Patients with EA, EGPA or HES
3. Provision of signed and dated written informed consent form prior to any mandatory study procedures, sampling and analysis.

Healthy donors:

1. Age between18 and 75 years healthy donors

Exclusion Criteria:

* Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

  1. Presence of other chronic pulmonary diseases including COPD
  2. Presence of other chronic immuno-mediated inflammatory diseases
  3. Treatment with oral prednisone or equivalent > 7.5 mg/day
  4. Treatment with long-acting depot corticosteroids in the last three months
  5. Use of immunosuppressive medications (cyclosporine A; azathioprine; methotrexate; mycophenolate mofetil)
  6. Receipt of live attenuated vaccines 30 days prior to the enrollment
  7. Acute upper or lower respiratory infections within 30 days prior to the date informed consent is obtained or during the screening/run-in period.
  8. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy
  9. Subjects who are pregnant or breastfeeding
  10. Current smoking
  11. Any clinically significant abnormal findings in physical examination, vital signs, hematology, or clinical chemistry during screening period, which in the opinion of the investigator may put the patient at risk of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study.
  12. Concurrent enrolment in another interventional or post-authorization safety study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Each subject should meet all of the inclusion criteria and none of the exclusion criteria for this study. Under no circumstances can there be exceptions to this rule.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary objective: first outcome measure | From the enrollment of the first patient at 20 months
  1) Proportion of circulating Siglec8+CD16-CD62Llow (iEos) and Siglec8+CD16-CD62Lbright (rEos) cells in bio- naïve, EGPA and HES patients
Primary objective: second outcome measure | From the enrollment of the first patient at 20 months
  2) Modification of the expression of CD62L on peripheral eosinophils upon in vitro stimulation with IL-5, IL-3, GM-CSF, IL-4, IL-13

SECONDARY OUTCOMES:
Secondary objective: first outcome measure | From the enrollment of the first patient at 18 months
  1) Proportion of circulating Siglec8+CD16-CD62Llow (iEos) cells in bio-naïve EA, EGPA, and HES patients
Secondary objective: second outcome measure | From the enrollment of the first patient at 18 months
  2) Correlation between Siglec8+CD16-CD62Llow (iEos) cells and disease-specific clinical scores in bio-naïve EGPA, HES and EA patients

OTHER OUTCOMES:
Explorative objective | From month 7 to month 20
  1) Modification of the proportion of CD62Llow and CD62Lbright among eosinophils obtained from EGPA and HES patients, upon in vitro coculture with mepolizumab and type 2 cytokines.

REFERENCES:
- [Background] Matucci A, Nencini F, Maggiore G, Chiccoli F, Accinno M, Vivarelli E, Bruno C, Locatello LG, Palomba A, Nucci E, Mecheri V, Perlato M, Rossi O, Parronchi P, Maggi E, Gallo O, Vultaggio A. High proportion of inflammatory CD62Llow eosinophils in blood and nasal polyps of severe asthma patients. Clin Exp Allergy. 2023 Jan;53(1):78-87. doi: 10.1111/cea.14153. Epub 2022 May 4. PMID 35490414
- [Background] Januskevicius A, Jurkeviciute E, Janulaityte I, Kalinauskaite-Zukauske V, Miliauskas S, Malakauskas K. Blood Eosinophils Subtypes and Their Survivability in Asthma Patients. Cells. 2020 May 18;9(5):1248. doi: 10.3390/cells9051248. PMID 32443594
- [Background] Xenakis JJ, Howard ED, Smith KM, Olbrich CL, Huang Y, Anketell D, Maldonado S, Cornwell EW, Spencer LA. Resident intestinal eosinophils constitutively express antigen presentation markers and include two phenotypically distinct subsets of eosinophils. Immunology. 2018 Jun;154(2):298-308. doi: 10.1111/imm.12885. Epub 2018 Jan 21. PMID 29281125
- [Background] Marichal T, Mesnil C, Bureau F. Homeostatic Eosinophils: Characteristics and Functions. Front Med (Lausanne). 2017 Jul 11;4:101. doi: 10.3389/fmed.2017.00101. eCollection 2017. PMID 28744457
- [Background] Mesnil C, Raulier S, Paulissen G, Xiao X, Birrell MA, Pirottin D, Janss T, Starkl P, Ramery E, Henket M, Schleich FN, Radermecker M, Thielemans K, Gillet L, Thiry M, Belvisi MG, Louis R, Desmet C, Marichal T, Bureau F. Lung-resident eosinophils represent a distinct regulatory eosinophil subset. J Clin Invest. 2016 Sep 1;126(9):3279-95. doi: 10.1172/JCI85664. Epub 2016 Aug 22. PMID 27548519
- [Background] Rosenberg HF, Dyer KD, Foster PS. Eosinophils: changing perspectives in health and disease. Nat Rev Immunol. 2013 Jan;13(1):9-22. doi: 10.1038/nri3341. Epub 2012 Nov 16. PMID 23154224